CLINICAL TRIAL: NCT03100305
Title: A Prospective Study of Amino Acids Profiles in Premature Infants Receiving Nutritional Support
Brief Title: Amino Acids Profiles in Premature Infants Receiving Nutritional Support
Status: Completed | Type: Observational
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Zhenjuan He, Deputy director of neonatal department, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: XH-17-001
Record Dates: First submitted 2017-02-21; First posted 2017-04-04 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Premature Infant
MeSH Terms: conditions — Premature Birth | interventions — Urination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Extremely preterm infants
  Interventions: Other: Collection of blood and urine
- Very preterm infants
  Interventions: Other: Collection of blood and urine
- Moderately preterm infants
  Interventions: Other: Collection of blood and urine
- Late preterm infants
  Interventions: Other: Collection of blood and urine

INTERVENTIONS:
Other: Collection of blood and urine — Collection of blood and urine before nutritional support, during total parenteral nutrition, during partial parenteral nutrition and during enteral nutrition

SUMMARY:
The aim of this study is to investigate the changes of amino acid metabolic profiles in different nutritional stages of preterm infants and determine the effects of nutritional intervention on the amino acid metabolic status of preterm infants.

ELIGIBILITY:
Inclusion Criteria:

Premature infants, and admitted to hospital within 24 hours after birth; Documentation of informed consent; In need of receiving parenteral nutrition after birth;

Exclusion Criteria:

Premature infants with a parenteral nutrition period of less than 3 days; Inborn error of metabolism; Chromosomal abnormalities or multiple malformations;

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Preterm infants who experience various nutritional stages including total parenteral nutrition, partial parenteral nutrition and enteral nutrition
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-03-20 (Actual)

PRIMARY OUTCOMES:
Amino acid profiles in blood | through the transition to enteral nutrition, an average of 1 month
  Amino acid levels in blood

SECONDARY OUTCOMES:
Weight | Until the corrected gestational age is 37 weeks or discharged
Height | Until the corrected gestational age is 37 weeks or discharged
Head circumference | Until the corrected gestational age is 37 weeks or discharged

CONTACTS AND LOCATIONS:
Overall Officials: Zhenjuan He, master, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No